CLINICAL TRIAL: NCT02880657
Title: Evaluation of SODB®, Associated With a Physical Training, in the Physical Condition Improvement in Healthy Subjects: Randomized Double-blind Study Versus Placebo
Brief Title: Evaluation of SODB® (Superoxide Dismutase by Bionov®) in the Physical Condition Improvement in Healthy Subjects
Acronym: MELORUN560
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bionov (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016-A00302-49
Record Dates: First submitted 2016-07-20; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
Keywords: superoxide dismutase; melon concentrate; oxidative stress; physical training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SODB®-physical training (Experimental): This arm receives daily two capsules of SODB® 40mg containing 560 UI of superoxide dismutase, associated with standardized physical training
  Interventions: Dietary Supplement: SODB®
- Placebo-physical training (Experimental): This arm receives daily two capsules of Placebo containing excipients only, associated with standardized physical training
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SODB® — Subjects are supplemented with SODB®, daily over 10 weeks. Each volunteer was seen for the 4 visits: - visit of pre-inclusion V1, - visit V2, so-called inclusion visit, - visit V3 after 4 weeks of physical training and - visit V3 after 8 weeks of physical training
  Arms: SODB®-physical training
Dietary Supplement: Placebo — Subjects are supplemented with Placebo, daily over 10 weeks. Each volunteer was seen for the 4 visits: - visit of pre-inclusion V1, - visit V2, so-called inclusion visit, - visit V3 after 4 weeks of physical training and - visit V3 after 8 weeks of physical training
  Arms: Placebo-physical training

SUMMARY:
The objective of this study is to evaluate the influence of a 10 weeks SODB® supplementation in physical condition improvements of healthy subjects, in comparison to a placebo.

DETAILED DESCRIPTION:
Beneficial experimental results have already been obtained with SODB®. That is why, the investigators expect several effects of SODB® here. Indeed, this clinical study could show that SODB® is able to improve physical conditions, and particularly at muscular and cardiac levels, by inducing a decrease in oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Ruffier score between 8 and 12
* 18.5 < Body Mass Index < 27 kg/m2
* stable weight (variation < 5% over the last 3 months)
* stable diet over the last 3 months
* normal biological exam
* arterial pressure < 140/90 mm Hg
* normal ECG
* no contraindication for running
* subject having given his free, informed and express consent
* subject affiliated with a social security insurance or beneficiary of such an insurance system
* time to go to the physical training twice per week

Exclusion Criteria:

* subject who do not understand the study
* > 5 cigarets per day
* slimming diet over the last 3 months
* contraindication for running or physical test
* subject who failed the Cooper test
* anormal ECG
* anormal biological results
* dyslipidemia
* under current statins treatment
* hypertension
* diabeta II
* chronic respiratory disease
* rheumatic disease
* orthopedic disease
* positive serology for hepatitis B, C or HIV
* under current corticoids treatment
* under current drugs (medicine or not)
* any allergy to utilized one of the compounds of the experimental or placebo product
* alcool > 36g/day
* consumption of drinks containing caffein, taurine, creatin, guarana, ginseng, ginkgo, biloba, etc
* consumption of drinks containing xanthic bases (> 0.5L/day)
* consumption of drinks containing plants (> 2L/day)
* consumption of grapefruit juice (> 0.5L/day)
* under current antioxidant treatment (and during last month)
* adult protected by the law
* any subject who participated to a clinical assay within the 3 months

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline physical condition at 10 weeks | Evaluation performed at inclusion day (V2) and after 5 weeks of treatment (V3) and 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by Ruffier test measurement

SECONDARY OUTCOMES:
Evaluation of cardiac frequence | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by measurements of cardiac frequence during a physical test
Evaluation of maximal aerobic vitesse | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by measurements of maximal aerobic vitesse during a physical test
Evaluation of maximal oxygen volume | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by measurements of maximal oxygen volume during a physical test
Evaluation of running time | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by measurements of running time during a physical test
Evaluation of running distance | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by measurements of running distance during a physical test
Evaluation of quality of fatigue | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by an auto scale (Prévost)
Evaluation of quality of life | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by an auto scale (SF36)
Evaluation of glucose blood level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by glucose measurements
Evaluation of insulin blood level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by insulin measurements
Evaluation of cholesterol level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by total and LDL-cholesterol measurements
Evaluation of triglycerides level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by triglycerides measurements
Evaluation of inflammation | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by CRP (C-reactive protein) measurements
Evaluation of ions modifications | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by ionogram measurements
Evaluation of creatinemia | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by creatinine measurements
Evaluation of lactate level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by lactate measurements
Evaluation of transaminases level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by transaminases measurements
Evaluation of cortisol level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by cortisol measurements
Evaluation of testosterone level | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by testosterone measurements

OTHER OUTCOMES:
Number of participants with treatment-related adverse events | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  All adverse events occured throughout the study analyzed in order to know the number of participants only with treatment-related adverse events
Description of oxidative marker modifications in blood | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by KRL (Kirial test) measurements
Description of antioxidant markers modifications in blood | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by antioxidant enzymes measurements
Description of Complete Blood Count modifications in blood | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
Description of serum protein modifications in blood | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by Serum Protein Electrophoresis measurements
Description of lymphocytes nature modifications in blood | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by lymphocytes families percent measurements
Description of Complement blood level modifications | Evaluation performed at inclusion day (V2) and after 10 weeks of treatment at the end of the study (V4)
  Evaluation performed by C3, C4 and CH50 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thalamas, Principal Investigator — CIC Hospital Purpan

IPD SHARING:
Plan to Share IPD: Undecided